CLINICAL TRIAL: NCT03873350
Title: The Effect of the Fermented Tea Beverage Kombucha on the Human Microflora: a Placebo-controlled Study
Brief Title: The Effect of the Fermented Tea Beverage Kombucha on the Oral and Gut Microflora
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Responsible Party: Principal Investigator, Åsa Håkansson, Assistant university lecturer at the Department of Food Technology, Lund University, Lund University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Kombucha study 2018
Record Dates: First submitted 2019-03-11; First posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Microbial Colonization
Keywords: Microbiota colonization kombucha bacteria yeast
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Intervention Model Description: The participants will be divided into three groups in which one is given living kombucha, one heat-sterilized kombucha (placebo group) and one regular tap water (control group).
Who Masked: Participant, Investigator
Masking Description: The participants will be masked, meaning they will not know if they are given living or sterilized kombucha. The control group consuming water will know that they are the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Living kombucha (Experimental)
  Interventions: Other: Consumption of kombucha
- Heat-sterilized kombucha (Placebo Comparator)
  Interventions: Other: Consumption of heat-sterilized kombucha
- Water (No Intervention)

INTERVENTIONS:
Other: Consumption of kombucha — The intervention performed in the study implies letting healthy individuals consume one bottle (33 cl) of living kombucha daily for three weeks.
  Arms: Living kombucha
Other: Consumption of heat-sterilized kombucha — The intervention performed in the study implies letting healthy individuals consume one bottle (33 cl) of heat-sterilized kombucha daily for three weeks.
  Arms: Heat-sterilized kombucha

SUMMARY:
The purpose of the project is to investigate if consumption of the fermented tea beverage kombucha has an effect on the gut and/or oral microbiota, and further if it depends on the content of living bacteria or is inherent even to sterilized kombucha. This will be studied by a clinical trial in which healthy individuals will be given living kombucha, sterilized kombucha or water. The participants will consume one bottle (33 cl) of their designated drink per day for 21 days. Fecal and saliva samples will be collected before, directly and ten days after the intervention. These will then be examined to see if there is a change in the micro flora due to the kombucha.

DETAILED DESCRIPTION:
The first part of the project focuses on studying the characteristics of the kombucha drink and microbial composition. The amount of living organisms in the drink will be determined by colony count. Apart from this, the culture will be studied to determine which organisms are present and which are dominant. After isolation of colonies found from culturing, Sanger sequencing will be used for characterization.

The second part, which consists of the human study, will be performed over a span of 3 weeks and the aim is that 60 persons take part. The participants should be healthy, and have no diagnosed gut or stomach problems, and be 18 years old or older. They will be divided into groups, where one will be given living kombucha, one group kombucha sterilized by boiling (placebo) and the final group plain water (control group). The participants will drink one bottle (33 cl) of their designated beverage daily for two weeks. Fecal and saliva samples will be collected before, directly after and 10 days after the intervention. The samples will then be studied by sequencing the present organisms, after having extracted them. The library preparation will be made using Illumina sequencing. If possible, the aim is also to re-isolate a species from the kombucha after the study.

The participants will be registered for the study as they sign a consent form. These forms will then be treated as confidential material, and therefore be kept locked away at the institution. Only participating researchers will have access to the forms.

The participants will store the samples collected during the study until they are handed in for analysis. The samples will be destroyed during analysis.

The sample size has been chosen to a maximum of 60 participants, due to economical boundaries, but mainly because similar studied have used even fewer participants. As this is a pilot study more is not necessary. The intervention time (three weeks) was determined by comparison to other studies, but also restricted by the time scope of the project.

ELIGIBILITY:
Inclusion Criteria:

* The participants should be above 18 years of age.
* The participants must live in proximity of Lund or Helsingborg to be able to leave samples collected.
* The participants should consider themselves healthy and have no gut or stomach problems.

Exclusion Criteria:

* The participants should not be diagnosed with any gut or stomach diseases or problems.
* The participants cannot consume any food with living microorganisms two weeks before, during of ten days after the intervention.
* Participants cannot use anti-microbial oral products during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-05-02 (Actual); Study Completion 2018-05-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome is a change in the composition of the gut of oral micro flora, measured by extraction and sequencing of genetic material in fecal and saliva samples. | Samples will be collected before, directly after and ten days after the end of the intervention.
  A library will be created using Illumina sequencing that will enable comparing the microbiological composition before and after the intervention.

SECONDARY OUTCOMES:
The secondary outcome of the study is to be able to re-isolate a species from the kombucha in the collected samples after the intervention. | Samples will be collected before, directly after and ten days after the intervention. The kombucha culture is studied before the intervention.
  The secondary outcome will be measured by comparing results from the sequencing of microbes in the collected human samples and from the kombucha drink itself.

CONTACTS AND LOCATIONS:
Locations (1):
- Lund University, Lund, Skåne County, Sweden

IPD SHARING:
Plan to Share IPD: No
No plan to share participant data.